CLINICAL TRIAL: NCT03513562
Title: Phase 2 Study of Venetoclax Added to Ibrutinib to Eliminate Ibrutinib Resistance Mutations in CLL
Brief Title: Venetoclax and Ibrutinib in Treating in Participants With Chronic Lymphocytic Leukemia and Ibrutinib Resistance Mutations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Kerry Rogers, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17387; NCI-2018-00410 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Ibrutinib Resistance
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, ibrutinib) (Experimental): Participants receive venetoclax PO daily on days 1-28 and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 or 24 courses in the absence of disease progression or unacceptable toxicity. Participants with MRD negativity after 12 or 24 courses discontinue treatment, while participants with MRD positivity continue treatment with venetoclax in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta

SUMMARY:
This phase II trial studies how well venetoclax and ibrutinib work in treating participants with chronic lymphocytic leukemia and have developed genetic mutations after previously being treated with ibrutinib. Venetoclax and ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if the addition of venetoclax to ibrutinib therapy can eliminate ibrutinib resistance mutations.

SECONDARY OBJECTIVES:

I. Determine the rate of minimal residual disease negative complete remission to combination ibrutinib and venetoclax therapy.

II. Determine progression-free survival after the addition of venetoclax to ibrutinib.

III. Determine overall survival after the addition of venetoclax to ibrutinib. IV. Describe the toxicity profile of venetoclax in combination with ibrutinib in this patient population.

EXPLORATORY OBJECTIVES I. Describe changes in variant allele frequency (VAF) of known ibrutinib resistance mutations after the addition of venetoclax.

II. Perform BH3 profiling and correlate with response to combination venetoclax and ibrutinib therapy.

III. Determine if increased expression of MCL-1 and BCL-XL is a potential mechanism of resistance to venetoclax when given in combination with ibrutinib.

IV. Determine potential mechanisms of resistance to ibrutinib and venetoclax combination treatment by whole exome and ribonucleic acid (RNA) sequencing.

OUTLINE: This is a dose escalation study of venetoclax.

Participants receive venetoclax orally (PO) daily on days 1-28 and ibrutinib PO once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 12 or 24 courses in the absence of disease progression or unacceptable toxicity. Participants with minimal residual disease (MRD) negativity after 12 or 24 courses discontinue treatment, while participants with MRD positivity continue treatment with venetoclax in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL) meeting criteria established in the World Health Organization (WHO) classification of hematologic disorders or International Workshop on Chronic Lymphocytic Leukemia (IWCLL)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Currently taking ibrutinib and first took ibrutinib > 3 months ago
* Presence of a known ibrutinib resistance mutation at ≥ 4% variant allele frequency OR < 4% with two separate measurements at least 4 weeks apart with increasing variant allele frequency
* Adequate bone marrow function independent of growth factor support at screening unless clearly due to marrow involvement by CLL and/or disease-related immune thrombocytopenia; if cytopenias are due to disease in the bone marrow any degree of cytopenias are allowed; patients with active uncontrolled autoimmune cytopenias are excluded
* Hemoglobin ≥ 8 g/dL
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3
* Platelets ≥ 40,000/mm^3
* Prothrombin time/partial thromboplastin time (PT/PTT) ≤ 1.5 x upper limit of normal (ULN) (unless receiving anticoagulation)
* Total bilirubin ≤ 1.5 x ULN (excepting Gilbert's syndrome)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ≤ ULN
* Creatinine clearance ≥ 40 mL/min/1.73m^2

  * Using 24-hour creatinine clearance or modified Cockcroft-Gault equation
* All patients must practice a highly effective method of birth control
* Able to take an absorb pill form oral medications
* Ability to understand and sign a written informed consent

Exclusion Criteria:

* Inability to continue taking ibrutinib for any reason
* Treatment with chemotherapy, immunotherapy, radiotherapy, targeted small molecule inhibitors, biologic agents, and/or an investigational therapy for 5 half-lives prior to first study dose of venetoclax; treatment with a biologic agent, such as a monoclonal antibody, for 30 days prior to study treatment; treatment with ibrutinib is allowed
* Need for anticoagulation with a vitamin K antagonist (warfarin); other anticoagulants and antiplatelet agents are allowed
* Treatment with a moderate or strong cytochrome P450 3A4 (CYP3A) inhibitor or inducer within 7 days prior to first dose of venetoclax or need for treatment with a strong CYP3A inhibitor or inducer during the period or the study; patients who have a need for treatment with a moderate CYP3A inhibitor or inducer during venetoclax dose escalation will also be excluded
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* History of lymphoma (Richter's syndrome) unless in complete remission > 2 years without relapse
* Known active involvement of the central nervous system by lymphoma or leukemia
* Known infection with the human immunodeficiency (HIV) virus
* A cardiovascular disability status of New York Heart Association Class ≥ 2, defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or angina pain
* Positive hepatitis serology:

  * Patients with positive serology for hepatitis B defined as positivity for hepatitis B virus surface antigen measurement (HBsAg) or anti-hepatitis B core total antibodies (antiHBc) may be considered for inclusion in the study on a case-by-case basis if they are hepatitis B viral deoxyribonucleic acid (DNA) negative and are willing to undergo ongoing hepatitis B virus (HBV) DNA testing by real-time polymerase chain reaction (PCR) monthly during the study
  * Patients with positive hepatitis B surface antigen (HBsAg) consistent with prior vaccination to HBV (i.e., hepatitis B immune status/anti-hepatitis B surface antibody [anti-HBs+], anti-HBc-) may participate
  * Patients suspected to have false positive serologic studies because of intravenous (IV) immunoglobulin administration are potentially eligible without need for further monitoring if they have negative PCR studies for viral DNA/RNA after discussion with the principal investigator
  * Patients with positive hepatitis C serology are excluded unless they have negative hepatitis C virus (HCV) ribonucleic acid (RNA) testing after receiving HCV-specific treatment and the case is discussed with the principal investigator
* Female patients who are pregnant, breast-feeding, or planning to become pregnant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of active malignancies other than chronic lymphocytic leukemia (CLL) within the past 3 years prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma or the cervix or breast
  * Basal cell or localized squamous cell carcinoma of the skin
  * Previous malignancy treated with curative therapy and not expected to relapse
* Inability to swallow capsules or tablets, or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption (malabsorption syndrome, resection of the small bowel, poorly controlled inflammatory bowel disease, etc.)
* Prior allogeneic stem cell transplant with day 0 < 12 months prior and/or with chronic graft versus host disease (GVHD) requiring current use of immunosuppression; patients with prior allogeneic stem cell transplant with day 0 > 12 months prior who do not require immunosuppression for GVHD will be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of mutation negative status after 12 courses of combination therapy of ibrutinib and venetoclax | Up to 3 years
  The rate of mutation negative status will be the percentage of patients who have negative testing for ibrutinib resistance mutations in the peripheral blood and bone marrow after 12 courses of combination ibrutinib and venetoclax treatment. Mutation negative status is defined as 1% variant allele frequency by the clinical grade test for mutation.

SECONDARY OUTCOMES:
Rate of minimal residual disease negative complete remission after 12 courses of venetoclax and ibrutinib | Up to 3 years
  Rate of minimal residual disease negative complete remission estimated with a 95% exact binomial at the response assessment after 12 courses of therapy.
Progression-free survival after adding venetoclax to ibrutinib | From start date of combination therapy up to 3 years
  Progression-free survival (PFS) calculated from the start date of combination therapy until the date of clinical disease progression by the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria or death from any cause, whichever occurs first. PFS described using the method of Kaplan-Meier. Median PFS reported with 95% confidence interval.
Overall survival after beginning venetoclax in combination with ibrutinib | From start date of combination therapy up to 3 years
  Overall survival (OS) calculated from the start date of combination therapy until the date of death from any cause, censoring patients alive at last follow-up. OS described using the method of Kaplan-Meier. Median OS reported with 95% confidence interval.
Discontinuation rate due to adverse events with combination venetoclax and ibrutinib treatment. | Up to 3 years
  Safety and tolerability of the combination regimen adverse events are summarized by type, severity and perceived attribution according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 with the exception of hematologic adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Rogers, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu